CLINICAL TRIAL: NCT02050048
Title: Perioperative Intravenous Administration of High Volume Lactated Ringer's Solution and the Risk of Post-Endoscopic Retrograde Cholangiopancreatography (ERCP) Pancreatitis
Brief Title: High Volume Lactated Ringer's Solution and Pancreatitis
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Study was closed prematurely due to low enrollment numbers.
Sponsor: Endeavor Health (Other)
Collaborators: Medical College of Wisconsin (Other); Allina Health System (Other); Wake Forest University Health Sciences (Other); University of Utah (Other)
Responsible Party: Principal Investigator, Rachel Pulido, Russelll Brown, M.D., Endeavor Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EH 13-130
Record Dates: First submitted 2014-01-27; First posted 2014-01-30 (Estimated); Results first posted 2016-04-29 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-08

CONDITIONS: Pancreatitis
Keywords: Pancreatitis; Endoscopic retrograde cholangiopancreatography; Cholangiopancreatography, Endoscopic Retrograde; ERCP; High Volume; Lactated Ringer; Intravenous Administration; Sphincterotomy, Endoscopic; Pancreas
MeSH Terms: conditions — Pancreatitis | interventions — Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High Volume Group (Intervention Arm) (Experimental): Patients will be randomized to receive intravenous Lactated Ringer's solution. In the high volume group (intervention arm), patients will receive fluids prior to, during, and after the completion of the procedure. Patients in the high volume group will receive fluids via infusion by the following weight based regimen:
  * initial bolus of LR prior to ERCP of 7.5 cc/kg over 1 hour
  * LR fluid infusion during the procedure at 5 cc/kg/hr
  * Post-procedure bolus of 20 cc/kg over 90 minutes
  Interventions: Other: Administration of Lactated Ringer's (LR) Solution
- Low Volume Group (Control Arm) (Active Comparator): Patients will be randomized to receive intravenous Lactated Ringer's solution. In the low volume group (control arm), patients will receive fluids at the start of the ERCP. The fluids will be administered via infusion at a rate of 1.5 cc/kg/hr. Fluids may be continued through the 90 minute post-procedure observation period.
  Interventions: Other: Administration of Lactated Ringer's (LR) Solution

INTERVENTIONS:
Other: Administration of Lactated Ringer's (LR) Solution — Patients will be randomized to low volume or high volume group. Patient in the low volume group will receive fluids via infusion at a rate of 1.5 cc/kg/hr. Fluid administration may be continued through the 90 minute post-procedure observation period. Patients in the high volume group will receive fluids via infusion by the following weight based regimen:
  * initial bolus of LR prior to ERCP of 7.5 cc/kg over 1 hour
  * LR fluid infusion during the procedure at 5 cc/kg/hr
  * Post-procedure bolus of 20 cc/kg over 90 minutes

SUMMARY:
The purpose of this study is to examine whether giving large amounts of intravenous (IV) fluids will reduce the risk of developing a complication known as post-ERCP pancreatitis (PEP). Pancreatitis is inflammation of the pancreas, and it is the most frequent serious complication of ERCP. Typically, a small amount of IV fluids are given during this procedure (~ 1 liter). We are testing whether using a larger amount of fluids (2 - 3 liters) will reduce the risk of PEP.

DETAILED DESCRIPTION:
This trial is designed as a phase II/III study. The phase II portion of the trial will be completed to establish safety and efficacy data prior to proceeding with a phase III study. The phase II trial will enroll 110 patients that are undergoing elective ERCP as outpatients. Following the phase II portion, if the data suggests that the intervention arm (high volume group) is safe, the investigators will begin enrolling patients who are undergoing ERCP in a more urgent setting as inpatients.

We plan on enrolling 1,400 consecutive high risk patients undergoing ERCP. We are assuming a baseline PEP risk of 9.2%. Fluid administration will be based on Ideal Body Weight (IBW) in order to standardize the aggressive fluid administration across all body weights and reduce the potential for adverse cardiopulmonary outcomes.

All participants will be monitored for 90 minutes following their procedure to assess the development of any adverse symptoms. Analysis by a data safety monitoring board (DSMB) will take place throughout the study. The DSMB is comprised of a panel of experts independent of NorthShore University HealthSystem.

ELIGIBILITY:
Inclusion Criteria:

Patients to be included in the study are those undergoing ERCP with the following:

* Clinical suspicion of sphincter of Oddi dysfunction
* History of post-ERCP pancreatitis (at least one episode)
* Pancreatic sphincterotomy
* Pre-cut (access) sphincterotomy
* Ampullectomy

Exclusion Criteria:

* Age < 18 years old
* Intrauterine pregnancy or breastfeeding mother
* Congestive heart failure
* Advanced/symptomatic coronary artery disease
* Known ascites
* Renal failure
* Active or recent gastrointestinal hemorrhage
* Acute pancreatitis within 72 hours prior to ERCP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russell Brown, MD, Principal Investigator — Endeavor Health; Mick Meiselman, MD, Study Director — Central Coast Gastroenterology; Zachary Smith, MD, Study Director — Medical College of Wisconsin
Locations (6):
- United States (6):
  - NorthShore University HealthSystem, Evanston, Illinois
  - NorthShore University HealthSystem, Highland Park, Illinois
  - Advocate Health Care, Skokie, Illinois
  - Minnesota Gastroenterology, Plymouth, Minnesota
  - University of Utah Health Care, Salt Lake City, Utah
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Background] Freeman ML, Nelson DB, Sherman S, Haber GB, Herman ME, Dorsher PJ, Moore JP, Fennerty MB, Ryan ME, Shaw MJ, Lande JD, Pheley AM. Complications of endoscopic biliary sphincterotomy. N Engl J Med. 1996 Sep 26;335(13):909-18. doi: 10.1056/NEJM199609263351301. PMID 8782497
- [Background] Elmunzer BJ, Scheiman JM, Lehman GA, Chak A, Mosler P, Higgins PD, Hayward RA, Romagnuolo J, Elta GH, Sherman S, Waljee AK, Repaka A, Atkinson MR, Cote GA, Kwon RS, McHenry L, Piraka CR, Wamsteker EJ, Watkins JL, Korsnes SJ, Schmidt SE, Turner SM, Nicholson S, Fogel EL; U.S. Cooperative for Outcomes Research in Endoscopy (USCORE). A randomized trial of rectal indomethacin to prevent post-ERCP pancreatitis. N Engl J Med. 2012 Apr 12;366(15):1414-22. doi: 10.1056/NEJMoa1111103. PMID 22494121
- [Background] Feurer ME, Adler DG. Post-ERCP pancreatitis: review of current preventive strategies. Curr Opin Gastroenterol. 2012 May;28(3):280-6. doi: 10.1097/MOG.0b013e3283528e68. PMID 22450899
- [Background] Choudhary A, Bechtold ML, Arif M, Szary NM, Puli SR, Othman MO, Pais WP, Antillon MR, Roy PK. Pancreatic stents for prophylaxis against post-ERCP pancreatitis: a meta-analysis and systematic review. Gastrointest Endosc. 2011 Feb;73(2):275-82. doi: 10.1016/j.gie.2010.10.039. PMID 21295641
- [Background] Fazel A, Quadri A, Catalano MF, Meyerson SM, Geenen JE. Does a pancreatic duct stent prevent post-ERCP pancreatitis? A prospective randomized study. Gastrointest Endosc. 2003 Mar;57(3):291-4. doi: 10.1067/mge.2003.124. PMID 12612504
- [Background] Wu BU, Hwang JQ, Gardner TH, Repas K, Delee R, Yu S, Smith B, Banks PA, Conwell DL. Lactated Ringer's solution reduces systemic inflammation compared with saline in patients with acute pancreatitis. Clin Gastroenterol Hepatol. 2011 Aug;9(8):710-717.e1. doi: 10.1016/j.cgh.2011.04.026. Epub 2011 May 12. PMID 21645639
- [Background] Gardner TB, Vege SS, Pearson RK, Chari ST. Fluid resuscitation in acute pancreatitis. Clin Gastroenterol Hepatol. 2008 Oct;6(10):1070-6. doi: 10.1016/j.cgh.2008.05.005. Epub 2008 Jul 10. PMID 18619920
- [Background] Warndorf MG, Kurtzman JT, Bartel MJ, Cox M, Mackenzie T, Robinson S, Burchard PR, Gordon SR, Gardner TB. Early fluid resuscitation reduces morbidity among patients with acute pancreatitis. Clin Gastroenterol Hepatol. 2011 Aug;9(8):705-9. doi: 10.1016/j.cgh.2011.03.032. Epub 2011 Apr 8. PMID 21554987
- [Background] Freeman ML, DiSario JA, Nelson DB, Fennerty MB, Lee JG, Bjorkman DJ, Overby CS, Aas J, Ryan ME, Bochna GS, Shaw MJ, Snady HW, Erickson RV, Moore JP, Roel JP. Risk factors for post-ERCP pancreatitis: a prospective, multicenter study. Gastrointest Endosc. 2001 Oct;54(4):425-34. doi: 10.1067/mge.2001.117550. PMID 11577302
- [Background] de-Madaria E, Soler-Sala G, Sanchez-Paya J, Lopez-Font I, Martinez J, Gomez-Escolar L, Sempere L, Sanchez-Fortun C, Perez-Mateo M. Influence of fluid therapy on the prognosis of acute pancreatitis: a prospective cohort study. Am J Gastroenterol. 2011 Oct;106(10):1843-50. doi: 10.1038/ajg.2011.236. Epub 2011 Aug 30. PMID 21876561
- [Background] Nasr JY, Papachristou GI. Early fluid resuscitation in acute pancreatitis: a lot more than just fluids. Clin Gastroenterol Hepatol. 2011 Aug;9(8):633-4. doi: 10.1016/j.cgh.2011.03.010. Epub 2011 Mar 21. No abstract available. PMID 21421079
- [Derived] Wu M, Jiang S, Lu X, Zhong Y, Song Y, Fan Z, Kang X. Aggressive hydration with lactated ringer solution in prevention of post-endoscopic retrograde cholangiopancreatography pancreatitis: A systematic review and meta-analysis. Medicine (Baltimore). 2021 Apr 23;100(16):e25598. doi: 10.1097/MD.0000000000025598. PMID 33879722

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Volume Group (Control Arm): In the low volume group (control arm), patients will receive fluids at the start of the ERCP. The fluids will be administered via infusion at a rate of 1.5 cc/kg/hr. Fluids may be continued through the 90 minute post-procedure observation period.
Period: Overall Study
Arm/Group | High Volume Group (Intervention Arm) | Low Volume Group (Control Arm)
Started | 14 | 12
Completed | 9 | 10
Not Completed | 5 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Death | 1 | 0
Not completed — Ineligible after ERCP | 4 | 1

BASELINE CHARACTERISTICS:
Population: Those randomized to either the high or low volume group
Groups:
- Low Volume Group (Control Arm): In the low volume group (control arm), patients will receive intravenous Lactated Ringer's solution at the start of the ERCP. The fluids will be administered via infusion at a rate of 1.5 cc/kg/hr. Fluids may be continued through the 90 minute post-procedure observation period.
- Total: Total of all reporting groups
Arm/Group | High Volume Group (Intervention Arm) | Low Volume Group (Control Arm) | Total
Number analyzed (Participants) | 14 | 12 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 8 | 17
  >=65 years | 5 | 4 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (11.9) | 55.7 (18.1) | 57.4 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 14 | 12 | 26
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.6 (6.6) | 25.6 (3.4) | 27.7 (5.5)
Creatinine [Mean (Standard Deviation); unit: mg/dL] | 0.83 (0.20) | 0.89 (0.22) | 0.86 (0.21)

OUTCOME MEASURES:

1. Primary Outcome: Development of Post-ERCP Pancreatitis
Description: Patients will be monitored after procedure to see if they develop abdominal pain. If so, serum amylase and lipase blood draws will be completed at least once every 24 hours following procedure to monitor the development of post-ERCP pancreatitis. If patients do not develop abdominal pain following the procedure, research staff will follow up with the patients 5 days and 29 days after the procedure to evaluate for the development of post-ERCP pancreatitis and other related or unrelated complications.
Time Frame: Assessed 90 minutes after procedure, 5 days after procedure, and 29 days after procedure
Measure: Number; unit: participants
Groups:
- Low Volume Group (Control Arm): Patients will be randomized to receive intravenous Lactated Ringer's solution. In the low volume group (control arm), patients will receive fluids at the start of the ERCP. The fluids will be administered via infusion at a rate of 1.5 cc/kg/hr. Fluid administration may be continued through the 90 minute post-procedure observation period.
Arm/Group | High Volume Group (Intervention Arm) | Low Volume Group (Control Arm)
Number analyzed (Participants) | 14 | 12
participants | 0 | 1

2. Secondary Outcome: Number of Participants With Adverse Events Related to Fluid Overload
Description: A portion of the study will assess whether there is a significant risk of adverse events related to fluid overload states in the high volume (HV) intervention arm. We anticipate the rate of adverse events in patients randomized to the HV arm to be small. By using more modest, weight based regimens, we aim to optimize benefit while eliminating overly aggressive fluid administration and causing undue harm.
Time Frame: Phase II portion (~1 year)
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | High Volume Group (Intervention Arm) | Low Volume Group (Control Arm)
Serious Adverse Events (participants affected / at risk) | 1/14 | 2/12
Other Adverse Events (participants affected / at risk) | 5/14 | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High Volume Group (Intervention Arm) (N=14) | Low Volume Group (Control Arm) (N=12)
Liver failure (Hepatobiliary disorders) | 1 | 0 — Due to pre-existing condition
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Lactic acidosis (General disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | High Volume Group (Intervention Arm) (N=14) | Low Volume Group (Control Arm) (N=12)
Abdominal pain (Gastrointestinal disorders) | 5 | 4
Fever (General disorders) | 0 | 3
Chills (General disorders) | 1 | 1
Edema (Blood and lymphatic system disorders) | 0 | 2

LIMITATIONS AND CAVEATS:
Due to low study enrollment, the study was terminated early. Beacuse only 26 subjects were enrolled, the study results may not be statistically significant.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes